CLINICAL TRIAL: NCT01917500
Title: Feasibility Study of Non-invasive and Continuous Measurement of Blood Pressure and Cardiac Output: Comparison to Non-invasive and Non-continuous Measurements
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: HeartBeat_V1.0
Record Dates: First submitted 2013-08-01; First posted 2013-08-06 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-08

CONDITIONS: Heart or Vascular Disease
Keywords: Continues non-invasive Blood pressure measurement; Continues non-invasive Cardiac Output measurement
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac ward 10 patients: 10 patients from the cardiac ward.

SUMMARY:
The objectives of this clinical trial is to validate a S/W application to compare the calculations of Hemodynamic parameters like Continuous blood pressure (BP) and Continuous cardiac output (CO). This Hemodynamic parameters are computed from Pulse Oximeter (PhotoPlethysmograph or PPG) signal with results obtained by NIBP intermittent measurements and Echocardiography. The first phase of the study will be done on 10 patients of the Cardiology dept.- Cardiac ICU, that have routine measurements of BP and CO using Echocardiography.

The HeartBeat system combines an FDA/CE approved watch-like Pulse Oximeter for acquiring the data and a Smartphone S/W application that serves as the Hemodynamic calculator. The S/W application performs POST-PROCESSING of the PhotoPlethismoGraphic (PPG) signal (Normally the PPG signal in Pulse Oximeters is used only to compute heart rate and SpO2). The raw data is transferred from the watch oximeter to the smartphone using a standard Bluetooth protocol.

The Post-processing uses wavelet signal processing to estimate and display certain Hemodynamic parameters like (Blood Pressure) BP and CO in a continuous and graphical way on a standard Android Smartphone. In addition to the standard heart rate and SpO2, the application displays the measured PPG signal and estimated continues BP and CO.

HeartBeat is the only device that can non-invasively estimate Continuous BP and its Cardiac Output component and the resistance component in a mobile wearable device. Differentiating between these 2 components can play a major role in helping the doctor to understand the effect of cardiovascular medications and Lifestyle interventions.

ELIGIBILITY:
Inclusion Criteria:

* Male and females
* Between the ages of 20-70 years old

Exclusion Criteria:

* Over 70 years old
* under 20 years old
* Supportive blood pressure
* Severe Sepsis
* Ventilated patients
* Supported by Amines
* Patients in state of Shock

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The trial will be conducted on a group of patients in the cardiac ward at the Rambam hospital. As long as they fall under the criteria, they will fit for the trial.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2013-08; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Cardiac Output | 1 month
  Patients in the cardiac department pass an echo-cardiograph procedure to measure their cardiac output. When it is done, we will attach our oximeter to the patient and using the application we will calculate Cardiac Output.
  We will compare between both measurements

SECONDARY OUTCOMES:
Blood Pressure | 1 month
  Patients in the cardiac department have their blood pressure often measured . When it is done, we will attach our oximeter to the patient and using the application we will calculate our blood pressure.
  We will compare between both measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Haifa, Israel